CLINICAL TRIAL: NCT00930865
Title: A Randomized, Open-Label, Parallel-group, Multiple-Dose Study to Evaluate the Potential Pharmacokinetic Interaction and Pharmacodynamic Effects on Renal Parameters of Bumetanide (1mg) and Dapagliflozin (10 mg) When Co-administered in Healthy Subjects
Brief Title: Study to Evaluate the Potential Pharmacokinetic Interaction and Pharmacodynamic Effects on Renal Parameters of Bumetanide (1mg) and Dapagliflozin (10 mg) When Co-administered in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB102-057
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bumetanide; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bumetanide (Active Comparator)
  Interventions: Drug: Bumetanide
- Dapagliflozin (Active Comparator)
  Interventions: Drug: Dapagliflozin
- Bumetanide + Dapagliflozin (Active Comparator)
  Interventions: Drug: Bumetanide; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Bumetanide — Tablets, Oral, 1 mg, Single Dose, 7 Days
  Other Names: Bumex
  Arms: Bumetanide; Bumetanide + Dapagliflozin
Drug: Dapagliflozin — Tablets, Oral, 10 mg. Single Dose, 7 Days
  Other Names: BMS-512148
  Arms: Bumetanide + Dapagliflozin; Dapagliflozin

SUMMARY:
To assess the potential pharmacokinetic (PK) interactions of bumetanide and dapagliflozin following multiple doses of 1 mg bumetanide and 10 mg dapagliflozin in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive. BMI = weight (kg)/ [height (m)]²
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized and men, ages 18 to 45

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Current smoker or recent (within 1 month) history of regular tobacco use
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Abnormal urinalysis at screening
* Glucosuria at screening
* Abnormal liver functions tests (ALT, AST or total bilirubin > 10 % ULN)
* Presence of edema on physical exam
* History of diabetes mellitus
* History of heart failure
* History of renal insufficiency
* History of chronic or recurrent UTI (defined as 3 occurrences per year) or UTI in the past 3 months
* Positive urine screen for drugs of abuse either at screening or before dosing
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
* History of allergy to SGLT2 inhibitors, bumetanide (or related compounds)
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)
* Prior exposure to dapagliflozin within 3 months of Day -1
* Exposure to any investigational drug or placebo within 4 weeks of Day -1
* Use of any prescription drugs within 4 weeks or over-the-counter acid controllers within 2 weeks prior to study drug administration
* Use of any other drugs, including over-the-counter medications within 1 week and herbal preparations, within 2 weeks prior to study drug administration
* Use of an oral, injectable or implantable hormonal contraceptive agent within 3 months of study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Exposure to the investigational drug will be measured to compare with and without the co-administration of other drugs | 24 hours post-dose on Day 8 and 15

SECONDARY OUTCOMES:
To assess the safety and tolerability of bumetanide and dapagliflozin following multiple oral doses of 1 mg bumetanide and 10 mg dapagliflozin, administered together, either simultaneously or after adaptation to either agent alone, in healthy subjects | during 14 days of dosing
Explore potential pharmacodynamic (serum/urine electrolytes) effects of bumetanide + dapagliflozin following multiple doses of 1 mg bumetanide + 10 mg dapagliflozin, administered together, either simultaneously or after adaptation to either agent alone | during 14 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- [Derived] Wilcox CS, Shen W, Boulton DW, Leslie BR, Griffen SC. Interaction Between the Sodium-Glucose-Linked Transporter 2 Inhibitor Dapagliflozin and the Loop Diuretic Bumetanide in Normal Human Subjects. J Am Heart Assoc. 2018 Feb 10;7(4):e007046. doi: 10.1161/JAHA.117.007046. PMID 29440005
- See also: MB102-057_redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3647&filename=MB102-057_redacted%20_CSR%20_synopsis.pdf